CLINICAL TRIAL: NCT01374464
Title: A Double Blind Randomised Control Trial Assessing Effects of Local Anaesthetic Concentration (0.5% vs 0.75%) and Volume (5mls vs 15mls) on the Respiratory Consequences of Ultrasound Guided Interscalene Brachial Plexus Nerve Block
Brief Title: Reducing Respiratory Side Effects of Interscalene Brachial Plexus Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Gillian Foxall, Royal Surrey County Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11/LO/0934
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Adverse Reaction to Peripheral Nerve- and Plexus-blocking Anesthetics
Keywords: Interscalene brachial plexus nerve block; Nerve block
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High Volume, High Concentration (Active Comparator)
  Interventions: Other: Interscalene brachial plexus block
- High Volume, Low Concentration (Active Comparator)
  Interventions: Other: Interscalene brachial plexus block
- Low Volume, High Concentration (Active Comparator)
  Interventions: Other: Interscalene brachial plexus block
- Low Volume, Low Concentration (Active Comparator)
  Interventions: Other: Interscalene brachial plexus block

INTERVENTIONS:
Other: Interscalene brachial plexus block — 4 different administrations of levobupivicaine will be applied:
  1. High Volume, High Concentration = 15mls of 0.75% levobupivicaine
  2. High Volume, Low Concentration = 15mls of 0.5% levobupivicaine
  3. Low Volume, High Concentration = 5mls of 0.75% levobupivicaine
  4. Low Volume, Low Concentration = 5mls of 0.5% levobupivicaine
  Other Names: Levobupivicaine; Chirocaine

SUMMARY:
Shoulder surgery is known to be extremely painful requiring high doses of opiate analgesics (morphine) to control pain. Morphine has numerous unwanted side effects including sedation, hallucinations and vomiting.

It is now standard procedure for patients undergoing shoulder surgery to have their pain controlled by means of an injection made around the nerves where they pass through the neck to supply the shoulder with sensation (similar to the numbing injections made by the dentist before a dental procedure). This injection is called a 'nerve block'.

Nerve blocks provide complete analgesia after shoulder surgery allowing clinicians to discharge patients home on the day of surgery, pain free and with no opiate side effects. However, a side effect of nerve blocks at this level is involvement of the phrenic nerve, which is anatomically close to the injection point. This may cause (temporary) paralysis of the diaphragm and in some cases, severe respiratory dysfunction.

Research shows that reducing either the volume or the concentration of the drug injected, can reduce the consequent respiratory dysfunction. However no study has compared both volume and concentration in parallel, to see which of these has the more significant effect in reducing respiratory dysfunction. Furthermore there has been no assessment of how these changes may affect the duration of analgesia received and patient coping after discharge.

The investigators propose to conduct a double blind randomised controlled trial at the Royal Surrey County Hospital, enrolling patients presenting for elective day case arthroscopic (key hole) surgery over a period of 6 months. Patients will receive one of four treatment allocations:

1. Low concentration-high volume of local anaesthetic
2. Low concentration-low volume of local anaesthetic
3. High concentration-high volume of local anaesthetic
4. High concentration-low volume of anaesthetic drug of local anaesthetic.

The aim of this study is to inform an optimum dosing regimen for patients in order to facilitate maximal pain relief and quality of recovery with minimum respiratory dysfunction.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing day case shoulder surgery that would normally be managed with a nerve block for post-operative pain relief will be considered eligible for the study. Inclusion criteria are detailed below

1. Age > 18 and < 80 years
2. American Society of Anaesthetists (ASA) grades I - III. (ASA grade determines how 'fit' a patient is for surgery, with 1 being a normal healthy patient and 5 being a moribund patient that is not expected to survive. 'Fitter' patients are being chosen as it is felt that severe associated illness may influence our results).
3. A composite pain score of 0 when assessed in the post anaesthetic care unit (PACU) at 30mins post-operatively. This will be required in order for the patient to be deemed to have an 'effective' nerve block and be entered into the study. Patients reporting pain at this point will be removed from the study and offered either a rescue brachial plexus block or alternative analgesia. (Published research by Riazi et al and by McNaught et al, indicates that 5mls of local anaesthetic solution is adequate for establishing an effective ISBPB in this immediate post-operative period).

Exclusion Criteria:

1. Significant respiratory disease including Chronic Obstructive Pulmonary Disease or unstable asthma
2. Renal or hepatic impairment
3. Allergy to local anaesthetic
4. Opiod tolerance (more then 30mg of morphine or its equivalent per day)
5. Body mass index > 40
6. Body weight < 56kg (due to potentially toxic doses of local anaesthetic drug if using higher volume of 0.75% concentration at below this weight)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-02 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Functional Vital Capacity post interscalene brachial plexus block | 30 minutes after waking in post operative care unit
  The functional vital capacity refers to the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Measuring FVC is done by spirometry.

SECONDARY OUTCOMES:
Quality of recovery from surgery | First 24 hours post-operatively
  By means of a quality of recovery questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Foxall, MBChB, MA, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust
Locations (1):
- Royal Surrey County Hospital, Guildford, Surrey, United Kingdom

REFERENCES:
- [Background] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Background] Riazi S, Carmichael N, Awad I, Holtby RM, McCartney CJ. Effect of local anaesthetic volume (20 vs 5 ml) on the efficacy and respiratory consequences of ultrasound-guided interscalene brachial plexus block. Br J Anaesth. 2008 Oct;101(4):549-56. doi: 10.1093/bja/aen229. Epub 2008 Aug 4. PMID 18682410
- [Background] McNaught A, Shastri U, Carmichael N, Awad IT, Columb M, Cheung J, Holtby RM, McCartney CJ. Ultrasound reduces the minimum effective local anaesthetic volume compared with peripheral nerve stimulation for interscalene block. Br J Anaesth. 2011 Jan;106(1):124-30. doi: 10.1093/bja/aeq306. Epub 2010 Nov 8. PMID 21059701
- [Background] al-Kaisy AA, Chan VW, Perlas A. Respiratory effects of low-dose bupivacaine interscalene block. Br J Anaesth. 1999 Feb;82(2):217-20. doi: 10.1093/bja/82.2.217. PMID 10364997